CLINICAL TRIAL: NCT06511154
Title: The Effect of Cognitive Exercise in Addition to Physical Exercise on Upper Extremity Functions, Balance and Cognitive Functions in Individuals With Multiple Sclerosis
Brief Title: The Effect of Cognitive Exercise on Upper Extremity Functions, Balance and Cognitive Functions in Multiple Sclerosis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara Yildirim Beyazıt University (Other)
Collaborators: Gulhane Training and Research Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 21.03.2024/03-641
Record Dates: First submitted 2024-07-16; First posted 2024-07-19 (Actual); Last update posted 2024-07-19 (Actual); Status verified 2024-07

CONDITIONS: Multiple Sclerosis
Keywords: Multiple Sclerosis; Cognitive Rehabilitation; LOTCA
MeSH Terms: conditions — Multiple Sclerosis | interventions — Cognitive Training

STUDY DESIGN:
Intervention Model Description: Parallel Assingment dual parallel group design
Who Masked: Outcomes Assessor
Masking Description: single (outcomes assessor) single (outcomes assessor) the evaulation of the patients will be carried out by a blinded investigator.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment group (Experimental): Patients in this group are the group in which a physiotherapy program consisting of cognitive rehabilitation and core-based upper extremity exercises will be applied.
  Interventions: Other: Cognitive Rehabilitation; Other: Core-based Upper Extremity Exercises
- Control group (Active Comparator): Patients in this group are the group in which a physiotherapy program consisting of core-based upper extremity exercises will be applied.
  Interventions: Other: Core-based Upper Extremity Exercises

INTERVENTIONS:
Other: Cognitive Rehabilitation — Cognitive rehabilitation is a treatment method used to regain or improve cognitive abilities.For the cognitive rehabilitation program, the Daily Exercise Package of the Norosoft Program, which mainly includes exercises to improve attention, information processing speed, verbal and visual memory functions, will be applied.
  Core-based Upper Extremity Exercises
  Breathing exercises, Core based stabilization and mobilization exercises Upper extremity exercises Coordination ve proprioception exercises
  Other Names: Core-based Upper Extremity Exercises
  Arms: Treatment group
Other: Core-based Upper Extremity Exercises — Breathing exercises, Core based stabilization and mobilization exercises Upper extremity exercises Coordination ve proprioception exercises

SUMMARY:
Multiple sclerosis (MS) is a chronic, progressive, demyelinating disease characterized by myelin sheath damage in the central nervous system that affects more than 2.5 million people worldwide and is more common in young adults aged 20-40 years, especially in women. Like physical impairments, cognitive impairments are a common clinical finding in individuals with MS, both in the early and late stages of the disease. Individuals with MS with cognitive impairment have more difficulty than those without cognitive impairment in participating in social and occupational activities, finding a job, working and performing routine household activities. It is also known that there is a high percentage of individuals with MS with upper extremity involvement in the early stages of the disease. Functional problems in the upper extremities lead to restriction of activity and participation in individuals with MS. Although it is stated that there is a high rate of upper extremity problems in individuals with MS, it is seen that they are not sufficiently understood and analyzed.

When the literature is examined; evidence-based studies examining the effect of cognitive exercise on motor functions in MS in addition to physical exercises are quite limited. In this context, the subject of this study is to examine the effect of cognitive rehabilitation on upper extremity functions, balance and cognitive functions in individuals with MS.

DETAILED DESCRIPTION:
Cognitive rehabilitation is a set of therapeutic approaches that aim to increase functional capacity by examining the relationship between brain and behavior in many areas of cognition such as attention, memory, concentration, reasoning, problem solving, judgment, motor planning and awareness, and the first goal of treatment is to minimize the loss of acquired neuro-cognitive function. Although cognitive rehabilitation programs have been shown to significantly slow down cognitive decline in studies on MS, rehabilitation studies are still in their infancy. In addition, the content and intensity of the rehabilitation program required to provide an effective result have not been clarified. Evidence-based studies examining the effect of cognitive exercise in addition to physical exercise on motor function in MS are also very limited. There are some studies investigating cognitive rehabilitation alone or physical rehabilitation, but to our knowledge, there are no studies investigating the superiority of cognitive rehabilitation over a classical physiotherapy program consisting of core-based upper extremity exercises. Therefore, more original and new studies are needed. Our study is important in this sense. The aim of this study was to show the effect of cognitive rehabilitation on upper extremity functions, balance and cognitive functions when it is applied in addition to physical rehabilitation in order to develop coping strategies by slowing down cognitive losses in individuals with MS and to ensure regeneration if possible. With the findings obtained as a result of the study, it is aimed to increase the quality of life of MS patients by increasing and developing cognitive rehabilitation programs in MS patients.

ELIGIBILITY:
Inclusion Criteria:

* Being between the ages of 18 and 65
* A definitive diagnosis of MS by a neurologist
* Having an Expanded Disability Status Scale (EDSS) score below 5.5
* No cognitive problems (Mini Mental Test score of 24 and above),
* Graduated from at least primary school
* No change in medical treatment in the last 6 months,
* Not having had an attack in the last 3 months and not using pulse steroid therapy
* Volunteering.

Exclusion Criteria:

* Having hearing and vision problems that prevent communication
* Having a neurological or psychiatric disease other than MS that causes cognitive impairment
* Pregnancy
* Oncological diseases
* Having other vestibular and orthopedic diseases that may affect balance
* Continue with a different exercise therapy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2024-05-13 (Actual); Primary Completion 2025-05-15 (Estimated); Study Completion 2025-06-15 (Estimated)

PRIMARY OUTCOMES:
Cognitive status | Change from baseline at 8 weeks treatment program after.
  Loewenstein Occupational Therapy Cognitive Assessment (LOTCA) was developed to assess basic cognitive abilities. It is a standardized method used between 6-70 years of age. This scale consists of 6 main sections and 26 subtests including orientation, visual perception, spatial perception, motor praxis, visual motor organization and thinking ability. It takes approximately 30-45 minutes to administer.
Upper extremity | Change from baseline at 8 weeks treatment program after.
  Manual Ability Measure-36: The scale includes 23 items with a wide range of difficulty that measure the functional level of patients.
  Nine Hole Peg Test: Evaluates unilateral fine motor skills in the upper extremity. It requires the participants to first insert the nine sticks one by one into the nine holes and then remove them as quickly as possible against the clock.
  Box and Block Test: It is used to measure hand gross skill performance.The patient is asked to transfer the maximum number of blocks, one at a time, from one compartment of a wooden box divided into two compartments to the other within 60 seconds.
  Jebsen - Taylor Hand Function Test: It is an standardized test used to measure fine and gross motor functions of the hand by simulating daily life activities. It consists of 7 subtests: writing, simulated number spinning, lifting small objects, simulated feeding, stacking, moving large light and heavy objects.

SECONDARY OUTCOMES:
Coordination | Change from baseline at 8 weeks treatment program after.
  The Finger to Nose Test is a practical test commonly used to assess coordination. The patient moves his/her arm from the fully extended position to the bent position, touches his/her finger to his/her nose and opens his/her arm again. The patient performs this movement consecutively. Another common one is that the patient touches his/her index finger to the clinician's index finger and then touches his/her own nose, this movement is repeated many times while the clinician continuously changes the position of his/her finger.
Balance | Change from baseline at 8 weeks treatment program after.
  Timed Up and Go Test: It is a method that evaluates the person's ability to move and requires both static and dynamic balance. In the test, the person is asked to get up from the chair, walk 3 meters at a safe and normal speed, turn, walk back and sit on the chair and the time is recorded in seconds. A shorter time indicates better balance and mobility. The starting position of the test is standardized.
  Berg Balance Scale: clinically evaluates functional balance and consists of 14 items related to functional tasks. These activities are ranked from the easiest to the most difficult. The items of the scale include activities requiring both dynamic and static balance. For each item, the level of competence in the activity is indicated by 5 points (0-4), with 0 being "unable" and 4 being "independent and safe". The maximum score is 56 points, with higher scores indicating better balance.
Fatigue | Change from baseline at 8 weeks treatment program after.
  Modified Fatigue Impact Scale: Will be used to measure fatigue. It is a modified version of the Fatigue Impact Scale based on items from interviews with MS patients about how fatigue affects their lives. It provides information about the effects of fatigue over the past four weeks in the physical (9 items), psychosocial (2 items) and cognitive (10 items) domains. The scale uses a 5-point Likert scale with 0 being 'Never' and 4 being 'Always'. An overall Modified Fatigue Impact Scale score of 38 or above is indicative of MS-related fatigue.
Position Sense | Change from baseline at 8 weeks treatment program after.
  Position Sense: Shoulder position sense will be measured for position sense measurement. Acumar dual digital inclinometer (Acu360, Acumar, Lafayette, USA) will be used to assess shoulder position sense. Before starting the tests, the test will be taught to the individuals both verbally and with practice in order to minimize the error rate. Shoulder abduction and flexion will be calculated at 30° and 60ᵒ. For both movements, the shoulder will start in neutral rotation position. Individuals will first be made to perform passive movement. After 3 seconds in this position, the shoulder will be brought to the neutral position. Afterwards, the individual will be asked to actively move the shoulder to the desired angle and movement and hold this position for 3 seconds with their eyes closed and express it aloud. Measurements will be repeated in both limbs (non-dominant and dominant) and a rest period of 60 seconds will be allowed between trials.

OTHER OUTCOMES:
Disability Status | Change from baseline at 8 weeks treatment program after.
  The Expanded Disability Status Scale (EDSS) will be used to determine the disability level of the patients. The scale consists of two parts. The functional systems section (pyramidal, cerebellar, brainstem, sensory, bowel and bladder, visual, cerebral or other) is graded from "0" no disability to "5" or "6" severe disability. The second section, assessing ambulation status, is based on the individual's functional system score and walking distance and is graded from "0" normal health to "10" death. The EDSS score of patients with mild-to-moderate (1-5.5) disabilities who will participate in the study will be determined by a specialist neurologist.
Cognitive Status | Change from baseline at 8 weeks treatment program after.
  Standardized Mini Mental Test (SMMT): It will be used to identify people who do not have cognitive problems, which is an inclusion criterion in the first stage. It is a short, easy-to-administer and standardized test that allows cognitive assessment in a short time and is used to determine the cognitive level globally. The test consists of five sub-headings: orientation, memory, attention, calculation, recall and language and is evaluated on a 30-point scale. Traditionally, scores between 24 and 30 are considered normal.

CONTACTS AND LOCATIONS:
Overall Officials: Emine İpek Halatcı, MSc, Principal Investigator — Ankara Yildirim Beyazıt University
Locations (1):
- Ankara Yıldırım Beyazıt University, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Indivudual participant data will be available to the responsible researcher.